CLINICAL TRIAL: NCT00911183
Title: Diffuse Large B Cell Non-Hodgkin's Lymphoma in the Vulnerable/Frail Elderly. A Multicentric Randomized Phase II Trial With Emphasis on Geriatric Assessment and Quality of Life
Brief Title: Diffuse Large B Cell Non-Hodgkin's Lymphoma in the Vulnerable/Frail Elderly. A Multicentric Randomized Phase II Trial
Acronym: FRAIL-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB-2008-25; IB-FRAIL06 (Other: Institut Bergonié); INCA-RECF0892 (Other: Institut National du Cancer); EUDRACT-2008-001506-16 (Other: EUDRACT)
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Results first posted 2022-06-14 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; pegfilgrastim; Rituximab; Cyclophosphamide; Prednisone; Vincristine

STUDY DESIGN:
Intervention Model Description: randomized non-comparative phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (R-COP regimen) (Experimental): Patients receive rituximab IV, cyclophosphamide IV, and vincristine sulfate IV on day 1. Patients also receive oral prednisone on days 1-5 and filgrastim subcutaneously (SC) on days 8-14 or pegfilgrastim SC on day 2. Treatment repeats every 21 days for at least 3 courses.
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: prednisone; Drug: vincristine sulfate
- Arm II (R-COPY regimen) (Experimental): Patients receive rituximab, cyclophosphamide, vincristine sulfate, prednisone, and filgrastim or pegfilgrastim as in arm I. Patients also receive liposome-encapsulated doxorubicin citrate IV on day 1. Treatment repeats every 21 days for at least 3 courses.
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: liposome-encapsulated doxorubicin citrate; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim — Given subcutaneously
Biological: pegfilgrastim — Given subcutaneously
Biological: rituximab — Given IV
Drug: cyclophosphamide — Given IV
Drug: liposome-encapsulated doxorubicin citrate — Given IV
  Arms: Arm II (R-COPY regimen)
Drug: prednisone — Given orally
Drug: vincristine sulfate — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, prednisone, and liposome-encapsulated doxorubicin citrate, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether rituximab and combination chemotherapy are more effective when given together with or without liposome-encapsulated doxorubicin citrate in treating older patients with diffuse large B-cell non-Hodgkin lymphoma.

PURPOSE: This randomized phase II trial is studying the side effects of giving rituximab together with cyclophosphamide, vincristine sulfate, and prednisone with or without liposome-encapsulated doxorubicin citrate and to see how well it works in treating older patients with stage II, stage III, or stage IV diffuse large B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the therapeutic efficacy of rituximab, cyclophosphamide, vincristine sulfate, and prednisone with vs without liposome-encapsulated doxorubicin citrate, in terms of complete remission rate at 6 months, in vulnerable or frail elderly patients with stage II, III, or IV diffuse large B-cell non-Hodgkin lymphoma.
* To assess the safety of these regimens in these patients.

Secondary

* To evaluate the progression-free survival, event-free survival, and overall survival rates at 6 and 24 months in patients treated with these regimens.
* To evaluate the overall response rate at 6 and 24 months in patients treated with these regimens.
* To evaluate the duration of complete remission in patients treated with these regimens.
* To evaluate the acute side effects (according to the International CTC scale) of these regimens in these patients.
* To evaluate the geriatric condition and quality of life of patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (R-COP regimen): Patients receive rituximab IV, cyclophosphamide IV, and vincristine sulfate IV on day 1. Patients also receive oral prednisone on days 1-5 and filgrastim subcutaneously (SC) on days 8-14 or pegfilgrastim SC on day 2. Treatment repeats every 21 days for at least 3 courses.
* Arm II (R-COPY regimen): Patients receive rituximab, cyclophosphamide, vincristine sulfate, prednisone, and filgrastim or pegfilgrastim as in arm I. Patients also receive liposome-encapsulated doxorubicin citrate IV on day 1. Treatment repeats every 21 days for at least 3 courses.

After 3 courses of R-COP or R-COPY, patients undergo evaluation. Patients with disease progression or a response of < 25% are removed from the study. Patients with a response of ≥ 25% receive 3 more courses of R-COP or R-COPY, followed by rituximab IV alone on day 1 of courses 7 and 8 in the absence of disease progression or unacceptable toxicity.

After the completion of chemotherapy, some patients may undergo radiotherapy.

Patients complete quality of life and geriatric assessment questionnaires at baseline and periodically during study treatment.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large B-cell non-Hodgkin lymphoma

  * Stage II, III, or IV disease (according to the WHO classification), including all morphological and clinical variants

    * No Burkitt-like lymphoma (presence of small cells in the bone marrow biopsy allowed)
  * CD20+ disease
* Has ≥ 1 measurable target lesion ≥ 1.1 cm (according to the International Workshop Criteria)
* Poor physiological status, as defined by ≥ 1 of the following criteria:

  * WHO performance status 3
  * Clinical evaluation and measurement of LVEF that would preclude doxorubicin administration (i.e., LVEF < 50%)
  * Creatinine clearance < 50 mL/min
  * Serum bilirubin > 30 μmol/L
  * Severe comorbidity that would preclude the use of CHOP chemotherapy
* Ineligible for standard R-CHOP therapy
* No cerebral or meningeal involvement

PATIENT CHARACTERISTICS:

* WHO performance status 0-3
* ANC > 750/mm^3
* Platelet count > 50,000/mm^3
* LVEF > 35%
* Able to receive either R-COP or R-COPY therapy
* No congestive heart failure, serious arrhythmia, or myocardial infarction within the past 6 months
* No other malignancy within the past 5 years except for adequately treated basal cell carcinoma of the skin or curatively treated carcinoma in situ of the cervix
* No active infection
* No active viral hepatitis B or C by serology
* No known HIV positivity
* No hypersensitivity to rituximab, any of its excipients, or to murine proteins
* No documented history of allergy to eggs or egg products
* No psychological, familial, sociological, or geographical condition that would preclude compliance with study treatment or follow-up schedule

PRIOR CONCURRENT THERAPY:

* No prior therapy for this cancer
* No prior anthracycline administration with a cumulative dose > 240 mg/m² of doxorubicin hydrochloride or > 400 mg/m² of epirubicin hydrochloride
* More than 30 days since prior participation in another clinical trial involving investigational drugs
* No other concurrent antineoplastic agents

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-12-02 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2015-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Soubeyran, MD, PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (R-COP Regimen) | Arm II (R-COPY Regimen)
Started | 47 | 20
Completed | 47 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (R-COP Regimen) | Arm II (R-COPY Regimen) | Total
Number analyzed (Participants) | 47 | 20 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.8 (4.2) | 81.1 (4.1) | 82.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 10 | 34
  Male | 23 | 10 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 47 | 20 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Complete Remission 6 Months After Randomization
Description: Complete remission [CR] is defined according to Cheson criteria. CR requires the following:
  1. Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities.
  2. All lymph nodes and nodal masses must have regressed to normal size. Previously involved nodes that were 1.1 to 1.5 cm in their greatest transverse diameter before treatment must have decreased to ≤1 cm in their greatest transverse diameter after treatment, or by more than 75% in the sum of the products of the greatest diameters (SPD).
  3. The spleen, if considered to be enlarged before therapy on the basis of a CT scan, must have regressed in size and must not be palpable on physical examination.
  4. If the bone marrow was involved by lymphoma before treatment, the infiltrate must be cleared on repeat bone marrow aspirate and biopsy of the same site.
Time Frame: 6 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (R-COP Regimen) | Arm II (R-COPY Regimen)
Number analyzed (Participants) | 47 | 20
Participants | 14 | 9

2. Primary Outcome: Number of Participants With Severe Toxicity
Description: Severe toxicity, defined as febrile neutropenia or toxic death. Febrile neutropenia is defined in the International CTC toxicity scale as "fever of unknown origin without clinically or microbiologically documented infection: neutrophils < 1.0 x 109/l and fever ≥ 38.5° C.
  Toxic death is defined as any death which occur during treatment (from day 1 of the first cycle of chemotherapy up to day 30 of the last cycle) and is not related to lymphoma.
Time Frame: 6 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (R-COP Regimen) | Arm II (R-COPY Regimen)
Number analyzed (Participants) | 47 | 20
Participants | 10 | 8

3. Secondary Outcome: Overall Survival Time
Description: OS is defined as the delay between the date of randomization and the date of death
Time Frame: from randomization, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (R-COP Regimen) | Arm II (R-COPY Regimen)
Number analyzed (Participants) | 47 | 20
months | 20.1 [10.4 to 25.4] | 25.4 [12.2 to NA] — the upper limit of 95%CI could not be estimated due to insufficient number of participants with events

4. Secondary Outcome: Progression-free Survival Time
Description: Delay between the date of randomization and the date of progression or death. Progression is defined according to the Cheson criteria.
Time Frame: from randomization, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (R-COP Regimen) | Arm II (R-COPY Regimen)
Number analyzed (Participants) | 47 | 20
months | 10.4 [5.4 to 25.9] | 18.0 [5.2 to NA] — he upper limit of 95%CI could not be estimated due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: up to 5 years after randomization
Description: Adverse events (other than serious) were not collected
Arm/Group | Arm I (R-COP Regimen) | Arm II (R-COPY Regimen)
All-Cause Mortality (participants affected / at risk) | 27/47 | 12/20
Serious Adverse Events (participants affected / at risk) | 46/47 | 20/20
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (R-COP Regimen) (N=47) | Arm II (R-COPY Regimen) (N=20)
Febrile aplasia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrythmia (Cardiac disorders) | 0 (0) | 1 (1)
Aurticular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
myocaridal infarct (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
other (Gastrointestinal disorders) | 1 (1) | 1 (1)
sigmoiditis (Gastrointestinal disorders) | 1 (1) | 0 (0)
asthenia (General disorders) | 1 (1) | 0 (0)
death (General disorders) | 1 (1) | 2 (2)
fever (General disorders) | 0 (0) | 1 (1)
general physical health deterioration (General disorders) | 2 (3) | 3 (3)
malaise (General disorders) | 1 (1) | 0 (0)
sudden death (General disorders) | 1 (1) | 0 (0)
biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Basterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Clotridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Enterobacter septicemia (Infections and infestations) | 0 (0) | 2 (2)
other (Infections and infestations) | 1 (1) | 0 (0)
pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 5 (5) | 1 (1)
virosis (Infections and infestations) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
femure fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
dehydratation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lymphomateous meningitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Accident cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
convulsion (Nervous system disorders) | 0 (0) | 1 (1)
other (Nervous system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatoid bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Distress respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes